CLINICAL TRIAL: NCT02543437
Title: The Effect of Large Diameter Head to Prevent Dislocation, and of 3 rd Generation Highly Crosslinked Polyethylene to Reduce Wear in Computer Assisted Total Hip Arthroplasty.
Brief Title: Large Head X3 Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stryker Japan K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJCR-OR-1002
Record Dates: First submitted 2015-08-10; First posted 2015-09-07 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-09

CONDITIONS: Degenerative Joint Disease
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trident Acetabular X3 Insert (Other): 28mm, 32mm and 36mm liner
  Interventions: Device: Trident Acetabular X3 Insert

INTERVENTIONS:
Device: Trident Acetabular X3 Insert

SUMMARY:
The purpose of this study is to explore the benefit of X3 polyethlene inserts with larger diameter heads used in the Japanese population. Range of Motion (ROM) and lift-off distance for both 28mm, 32mm and 36mm in patients will be examined intraoperatively by using the Stryker computerized tomography (CT) based Navigation system. Another aspect of this study is to observe wear resistance performance of X3 over historical liner existing highly crosslinked polyethylene.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who is a candidate for primary total hip arthroplasty (THA) with cementless acetabular and femoral components.
2. Patient who has diagnosis of degenerative joint disease and no bacterial infectious disease.
3. Patient whose age is 20 or over.
4. Patient who signed an Institutional Review Board (IRB)-approved, study specific Informed Patient Consent Form.
5. Patient who is willing and able to comply with postoperative scheduled evaluations.

Exclusion Criteria:

1. Patient who has a bacterial infectious disease or has a high risk of a bacterial infection.
2. Patient who requires revision surgery of a previously implanted total hip arthroplasty.
3. Patient who is morbidly obese, defined as having a Body Mass Index (BMI) > 45.
4. Patient who is or may be pregnant female.
5. Patient who has a neuromuscular or neurosensory deficiency, which limits ability to evaluate the safety and efficacy of the device.
6. Patient with diagnosed systemic disease (i.e. Paget's disease, renal osteodystrophy).
7. Patient who is immunologically suppressed or receiving chronic steroids.
8. Patient who is judged ineligible with specific reason by primary doctor.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2019-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Nagoya Kyoritsu Hospital, Nagoya, Aichi-ken
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Kyowakai Hospital., Suita, Osaka
  - Osaka City General Hospital., Osaka

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 117 participants / 120 hips enrolled in study.
Groups:
- Trident Acetabular X3 Insert: Trident Acetabular X3 Insert 28mm, 32mm and 36mm liner
Period: Overall Study
Arm/Group | Trident Acetabular X3 Insert
Started | 117
Completed | 117
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- X3 Liner: X3 28mm, 32mm and 36mm liner
  Trident Acetabular X3 Insert
Arm/Group | X3 Liner
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 17
Region of Enrollment [Number; unit: participants]
  Japan | 117

OUTCOME MEASURES:

1. Primary Outcome: Range of Motion(ROM) (Degree)
Description: Measure and compare the ROM using femoral head trials of 36mm- and 28mm-diameter during intraoperative confirmation.
Time Frame: Intraoperative
Population: Comparison between 28mm liner and 36mm line. Participants with available data : 119 hips in 117 participants.
Measure: Mean (Standard Deviation); unit: Degree
Units Other Than Participants: Hips
Arm/Group | X3 Liner
Number analyzed (Participants) | 117
Number analyzed (Hips) | 119
Degree
  Maximam Flexion | 2.6 (4.5)
  Maximam Extension | 2.6 (4.7)
  Maximam Abduction | 2.6 (4.5)

2. Primary Outcome: Lift Off Distance in Dislocation Maneuver(mm)
Description: Measure and compare the lift off distance in dislocation maneuver using femoral head trials of 36mm- and 28mm-diameter during intraoperative confirmation.
Time Frame: Intraoperative
Population: participants with available data : 100 hips in 100 participants.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Hips
Arm/Group | X3 Liner
Number analyzed (Participants) | 100
Number analyzed (Hips) | 100
mm
  Cup inclination | -0.2 (3.5)
  Cup anteversion | 1.4 (5.3)
  Stem anteversion | -1.2 (6.4)

3. Secondary Outcome: Wear Rate(%)
Description: Retrospective comparison of the wear amount over time between X3 liner and Crossfire insert.
Time Frame: 1 year, 2 years, 3 years and 5 years after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse Events were not collected.
Arm/Group | X3 Liner
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No